CLINICAL TRIAL: NCT00989573
Title: A Multinational, Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-finding and Confirmatory Trial of OPC-6535 in Patients With Active Crohn's Disease
Brief Title: A Dose-finding and Confirmatory Trial of OPC-6535 in Patients With Active Crohn's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 197-08-001; JapicCTI090915
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — tetomilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): oral administration of placebo once-daily for 8weeks
  Interventions: Drug: Placebo
- OPC-6535 25 mg (Experimental): oral administration of OPC-6535 25 mg once-daily for 8 weeks
  Interventions: Drug: OPC-6535
- OPC-6535 50 mg (Experimental): oral administration of OPC-6535 50mg once-daily for 8 weeks
  Interventions: Drug: OPC-6535

INTERVENTIONS:
Drug: Placebo — oral administration of placebo once-daily for 8 weeks
  Arms: Placebo
Drug: OPC-6535 — oral administration of OPC-6535 25 mg once-daily for 8 weeks
  Arms: OPC-6535 25 mg
Drug: OPC-6535 — oral administration of OPC-6535 50 mg once-daily for 8 weeks
  Arms: OPC-6535 50 mg

SUMMARY:
The purpose of this study is to verify the safety and efficacy of OPC-6535 and determine the optimal dose by once-daily oral administration of OPC-6535 at 25 or 50 mg or placebo for 8 weeks in combination with base treatment (either a fixed oral dose of 5-aminosalicylic acid [5-ASA] or a fixed oral dose of 5-ASA plus enteral nutrition) in 180 patients with active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Primary lesion in either small intestine or large intestine
* C-reactive protein (CRP) level above the upper limit of the normal range
* Patients who have been receiving a 5-ASA formulation (oral mesalazine) at a fixed dose of 2.25 g/day or higher (not exceeding the approved dose) and at a fixed dosing regimen
* Patients who have not received enteral nutrition or who have been receiving enteral nutrition at a fixed intake of 1200 kcal/day or less

Exclusion Criteria:

* Patients with an uncontrolled external fistula (including anal fistula)
* Patients with a history of total proctocolectomy or subtotal colectomy
* Patients with short bowel syndrome
* Patients with an artificial anus
* Patients with serious infectious disease (intra-abdominal abscess, etc)
* Patients with malignant tumor
* Female patients who are pregnant, lactating, or possibly pregnant, or who wish to become pregnant during the trial period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 191 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Chair — OPCJ
Locations (11):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region
- South Korea (4):
  - Busan
  - Daegu
  - Gyronggi-do
  - Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-6535 25 mg: Oral administration of OPC-6535 25 mg once daily for 8 weeks (started from 12.5 mg for the first week and the dose was titrated to 25 mg from the second week)
- OPC-6535 50 mg: Oral administration of OPC-6535 50mg once daily for 8 weeks (started from 12.5 mg for the first week and the dose was titrated to 25 mg from the second week, with further titration to 50 mg from the third week)
- Placebo: Oral administration of placebo once daily for 8 weeks
Period: Overall Study
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Started | 65 | 63 | 63
Completed | 52 | 41 | 55
Not Completed | 13 | 22 | 8
Not completed — Adverse Event | 8 | 12 | 4
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 7 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set comprised all subjects who received at least one dose of investigational medicinal product (IMP) and for whom postdosing efficacy data were obtained.
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo | Total
Number analyzed (Participants) | 64 | 63 | 61 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (10.2) | 30.5 (10.3) | 32.2 (9.5) | 31.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 23 | 53
  Male | 44 | 53 | 38 | 135
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 24 | 22 | 23 | 69
  Japan | 40 | 41 | 38 | 119

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement Rate (Number of Subjects Showing Clinical Improvement / Number of Subjects Evaluated × 100) After 8 Weeks of IMP Administration
Description: Definition of clinical improvement: Total Crohn's Disease Activity Index (CDAI) score improved by at least 70 points from the baseline score or to below 150 (CDAI < 150: remission, CDAI > 450: severe disease)
Time Frame: Week 8
Population: Full analysis set comprised all subjects who received at least one dose of IMP and for whom postdosing efficacy data were obtained.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 64 | 62 | 61
percentage of participants | 31.3 [20.2 to 44.1] | 21.0 [11.7 to 33.2] | 29.5 [18.5 to 42.6]

2. Secondary Outcome: Clinical Improvement Rate After 4 Weeks of IMP Administration
Description: Definition of clinical improvement: CDAI score improved by at least 70 points from the baseline score or to below 150 (CDAI < 150: remission, CDAI > 450: severe disease)
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 63 | 62 | 60
percentage of participants | 30.2 [19.2 to 43.0] | 16.1 [8.0 to 27.7] | 28.3 [17.5 to 41.4]

3. Secondary Outcome: Remission Rate (Number of Subjects Showing Remission / Number of Subjects Evaluated x 100) After 4 and 8 Weeks of IMP Administration
Description: Definition of remission: Total CDAI score improved to below 150
Time Frame: Weeks 4 and 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 64 | 63 | 61
percentage of participants
  Week 4: number analyzed (Participants) | 63 | 62 | 60
  Week 4 | 15.9 [7.9 to 27.3] | 6.5 [1.8 to 15.7] | 10.0 [3.8 to 20.5]
  Week 8: number analyzed (Participants) | 64 | 62 | 61
  Week 8 | 20.3 [11.3 to 32.2] | 11.3 [4.7 to 21.9] | 18.0 [9.4 to 30.0]

4. Secondary Outcome: Mean Change From Baseline in C-reactive Protein (CRP) Level After 4 and 8 Weeks of IMP Administration
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 64 | 63 | 61
mg/dL
  Week 4: number analyzed (Participants) | 63 | 63 | 60
  Week 4 | -0.19 (1.25) | -0.16 (2.35) | 0.24 (1.58)
  Week 8 | -0.03 (1.92) | -0.36 (2.19) | 0.34 (1.54)

ADVERSE EVENTS:
Time Frame: From the start of IMP administration up to 3 weeks after the end of the trial
Description: Adverse events (AEs) occurring after IMP administration were included in assessment of AEs.
  The safety analysis population comprised subjects who received at least one dose of IMP.
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 8/65 | 10/63 | 4/63
Other Adverse Events (participants affected / at risk) | 39/65 | 35/63 | 33/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-6535 25 mg (N=65) | OPC-6535 50 mg (N=63) | Placebo (N=63)
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 6 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 1 | 0
Pulmonary tuberculoma (Infections and infestations) | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-6535 25 mg (N=65) | OPC-6535 50 mg (N=63) | Placebo (N=63)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 2 | 0
Abdominal pain (Cardiac disorders) | 4 | 1 | 1
Abdominal pain upper (Cardiac disorders) | 1 | 0 | 3
Crohn's disease (Cardiac disorders) | 4 | 5 | 7
Dental caries (Cardiac disorders) | 1 | 2 | 0
Nausea (Cardiac disorders) | 9 | 10 | 3
Stomatitis (Cardiac disorders) | 0 | 2 | 2
Vomiting (Cardiac disorders) | 2 | 3 | 2
Malaise (General disorders) | 3 | 1 | 1
Pyrexia (General disorders) | 2 | 0 | 2
Influenza (Infections and infestations) | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 3 | 7
Parotitis (Infections and infestations) | 0 | 0 | 2
Blood triglycerides increased (Investigations) | 2 | 1 | 0
Blood urine present (Investigations) | 3 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 9 | 8 | 4
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No